CLINICAL TRIAL: NCT02898935
Title: Improvement of the Accuracy of Spatial Representation of Invasive Exploratory Electrodes in Focal Epilepsy
Acronym: ELEC3D
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MCX_2015_32
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-01

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Reconstruction software allows visualization of cortical structure in 3 dimensions, showing on a single picture the position of all the electrodes. The EEG signal of each recording plot of the electrode is analyzed and compared with the underlying brain structure reconstructed by the software. It is therefore possible to visualize 1) ictogenic and epileptogenic areas using neurophysiological stereoelectroencephalography (SEEG) data and 2) adjacent functional cortical areas with functional imaging and SEEG. Software makes it possible to determine the links between these areas. This study aims to show that using these software is an asset in surgical decision and in the choice of surgical strategy.

Each patient has presurgical evaluation (usual care), including morphologic and (if necessary) functional MRI, EEG and SEEG. In this study, software will be used to analyze the processed data (FSL software, FMRIB laboratory, Oxford University and BrainVisa/Anatomist. The surgical decision will be taken according to the usual staff procedures, based on the usual examination results. After the decision making process, the staff will be asked to reconsider the surgical decision, according to the analysis provided by the software. The discrepancies between the decisions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* children aged 18 months to 17 years old
* drug resistant focal epilepsy
* scheduled for deep brain electrodes exploration to assess surgical indication

Exclusion Criteria:

* contraindication to anesthesia or surgery
* refusal (of parents or child) to participate in the study
* no health insurance coverage

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with drug resistant focal epilepsy, potential candidates for surgery, scheduled for deep brain electrodes exploration.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
number of patients for whom surgical strategy would change if using the software | 1 day
  change in medical strategy includes surgery indication, resection volume, topography of resection area

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CHIPAUX, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France